CLINICAL TRIAL: NCT03632226
Title: Evaluation of a Novel PET Radioligand to Image OGA
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 160105; 16-M-0105
Record Dates: First submitted 2018-08-14; First posted 2018-08-15 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06-25

CONDITIONS: Pharmacokinetics; Adult
Keywords: PET Imaging; Neurodegeneration
MeSH Terms: conditions — Nerve Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Healthy Volunteers
  Interventions: Drug: 18F-OGA-1

INTERVENTIONS:
Drug: 18F-OGA-1

SUMMARY:
Background:

O-GlcNAcase (OGA) is a brain enzyme. It may play a role in brain disorders like Alzheimer s disease. Researchers want to see if a new drug can be used with positron emission tomography (PET) scans to show OGA better. Researchers want to learn more about how it acts in healthy people.

Objectives:

To test if the new drug [18F]OGA-1 can measure its receptor. To determine whether the same results occur when scanning a person twice.

Eligibility:

Healthy adults age 18 and older who are already enrolled in a separate protocol.

Design:

Some participants will have 1 whole-body PET scan during one 4-hour visit to the clinic. Some will have 2-3 brain scans (PET and MRI) over 2-3 days.

For the PET scan, a needle will guide a thin plastic tube (IV catheter) into an arm vein. A small amount of radioactive chemical will be injected through the catheter. The needle will be removed. Only the catheter will be left in the vein.

Another IV catheter may be placed to draw blood.

Blood pressure, heart rate, and breathing rate will be measured. Participants will have an electrocardiogram.

Participants will lie on a bed that slides in and out of the donut-shaped scanner.

The scan will last 2-3 hours.

For brain PET scan, participants will wear a plastic mask to keep their head still.

For magnetic resonance imaging (MRI) scan, participants will lie on a table. The table slides in and out of the MRI scanner. This is a metal cylinder in a strong magnetic field. Participants will be in the scanner up to 1 hour.

DETAILED DESCRIPTION:
Objective:

Tau, a microtubule associated protein, regulates axonal structure and function within neurons of the brain. Neurofibrillary tangles contain hyper-phosphorylated, insoluble tau protein and are a hallmark of Alzheimer s disease (AD) and other tauopathies. Hyperphosphorylation of tau is required for its aggregation into tangles. One novel strategy to decrease the phosphorylation of tau is to increase the number of sugar molecules attached to tau, with the overly simple mechanism that the presence of the sugar molecules physically blocks phosphorylation. In this case, the sugar molecule is N-acetyl-Beta-D-glucosamine (GlcNAc), and increased glycosylation is achieved by inhibiting the enzyme (OGA) that removes these residues.

In collaboration with Eli Lilly, our laboratory recently developed (18F)OGA-1, a novel PET ligand to image the hydrolase OGA (O-GlcNAcase). Initial PET scans in monkey demonstrated that (18F)OGA-1 is a promising ligand.

This protocol is a first-in-human evaluation of (18F)OGA-1 and has four phases:

1. Phase 1: whole body imaging of one (1) subject with a low injection activity of approximately 2 mCi to confirm that no organ has prominently high uptake of (18F)OGA-1;
2. Phase 2: kinetic brain imaging in ten (10) subjects with up to 5 mCi injection to quantify OGA in brain relative to concurrent measurement of the parent radioligand in arterial plasma and venous plasma;
3. Phase 3: if (18F)OGA-1 is successful in Phase 2 in the first couple of subjects, we will estimate the radiation-absorbed doses by performing whole body imaging on a total of eight (8) subjects, with 5 mCi injection;
4. Phase 4: test-retest analysis in twelve (12) subjects, of brain binding relative to concurrent measurement of the parent radioligand in arterial plasma (5 mCi per scan) and venous plasma.

Thus, a total of 9 for whole body imaging and 22 for brain imaging

Study Population:

Healthy adult female and male volunteers (n= 22, ages greater than or equal to 18) will undergo brain imaging. An additional nine healthy volunteers will undergo whole body dosimetry analysis, for a total of 31 healthy volunteers.

Design:

For quantification of (18F)OGA-1, 22 healthy controls will undergo brain PET imaging using [18F]OGA-1 an arterial line, and venous line. Of this group of 22 healthy controls having brain PET imaging, twelve of them will have a test-retest scan. Nine additional subjects will have a whole body PET scan for dosimetry. For dosimetry, no arterial line will be used.

<TAB>

Outcome Measures:

To assess quantitation of OGA with (18F)GA-1, we will primarily use two outcome measures, namely the identifiability and time stability of distribution volume (VT) calculated with compartmental modeling. In the test-retest study, we will calculate the retest variability. We will assess whole-body biodistribution and dosimetry of (18F)OGA-1 by calculating doses to organs and the effective dose to the body as a whole.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age greater than or equal to 18.
* Able to give written informed consent.
* Medically and psychiatrically healthy.
* Enrolled in 01-M-0254 The Evaluation of Participants with Mood and Anxiety Disorders and Healthy Volunteers (PI: Dr. Carlos Zarate).

EXCLUSION CRITERIA:

* Any current Axis I diagnosis, based on interview and self-reporting performed under screening protocol 01-M-0254.
* Clinically significant laboratory abnormalities, based on tests performed under screening protocol 01-M-0254 that may include: CBC, acute care panel, hepatic panel, mineral panel, UA, urine drug screen, urine HCG (females), vitamin B12, folate, lipid panel, hepatitis panel (A, B, C), RPR, total protein, hs-CRP, uric acid, CK, LDH, thyroid panel, PT/PTT, and EKG.
* Positive HIV test.
* Unable to have an MRI scan.
* History of medical or neurologic illness / injury with the potential to affect study data interpretation.
* Recent exposure to radiation related to research (i.e. PET from other research) that, when combined with this study, would be above the allowable limits.
* Inability to lie flat on camera bed for at least two hours.
* Pregnancy or breastfeeding.
* Current drug/alcohol abuse or dependence.
* NIMH employees/staff and their immediate family members will be excluded from the study per NIMH policy.

Exclusion criteria for the dosimetry subjects are the same as reported above, with the exception of MRI contraindications, because an MRI will not be performed in these subjects.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2016-05-02; Primary Completion 2019-06-25 (Actual); Study Completion 2019-06-25 (Actual)

PRIMARY OUTCOMES:
The indentifiability and time stability of the distribution volume calculated with compartmental modeling of [F18 OGA-1]. In the test-retest study the retest variability will be calculated. | Ongoing

SECONDARY OUTCOMES:
Whole-body distribution and dosimetry of [18F]OGA-1 | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Innis, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States